CLINICAL TRIAL: NCT06276309
Title: Protein Molecular Characteristics and Prognosis of Cervical Neuroendocrine Tumors
Status: Recruiting | Type: Observational
Sponsor: Fujian Maternity and Child Health Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NECC2401
Record Dates: First submitted 2024-02-07; First posted 2024-02-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Neuroendocrine Neoplasm; China; Women; Cervical Cancer; Cervical Lesion
MeSH Terms: conditions — Neuroendocrine Tumors; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Paraffin samples collected from 100 cases of cervical neuroendocrine tumors were identified, processed and segmtioned, and protein concentration and proteome were determined to establish the molecular characteristics and prognostic targets of cervical neuroendocrine tumors.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The clinical diagnosis and treatment data of 300 cases of cervical neuroendocrine tumors were collected, including age, preoperative biopsy pathology results, postoperative histopathological results, TCT results, and colposcopy biopsy pathology results. At the same time, paraffin tissue specimens (remaining specimens after pathological diagnosis) from 100 cases of cervical neuroendocrine tumors from multiple centers across the country were collected to establish a cervical neuroendocrine tumor data follow-up database. Protein concentration and omics analysis were performed on the data results, to evaluate the molecular characteristics and prognosis of cervical neuroendocrine tumor proteins, and to preliminarily explore its clinical application value.

DETAILED DESCRIPTION:
1. The clinical diagnosis and treatment data of 300 cases of cervical neuroendocrine tumors were used for prognostic analysis.

(1) The diagnosis and treatment information of cervical neuroendocrine carcinoma in multiple hospitals was collected, including clinical and medical data such as age, preoperative HPV genotyping, preoperative biopsy pathological results, postoperative histopathological results, FIGO staging, prognosis and survival information, and follow-up of patients.

2. Protein and other omics analysis was performed on paraffin tissues of 100 cases of cervical neuroendocrine tumors Paraffin samples collected from 100 cases of cervical neuroendocrine tumors were identified, processed and segmtioned, and protein concentration and proteome were determined to establish the molecular characteristics and prognostic targets of cervical neuroendocrine tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with cervical neuroendocrine carcinoma by histopathology
2. Clinical data were complete

Exclusion Criteria:

1. Patients who are not being treated in our hospital
2. Patients with lack of follow-up data, unable to obtain survival information
3. Patients call to refuse to participate in this project
4. The quality of paraffin specimens can not meet the requirements of proteome concentration determination

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All 300 patients were diagnosed with cervical neuroendocrine carcinoma by histopathology
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
mortality rate | Among patients with cervical neuroendocrine carcinoma, the mortality rate within 3 years following surgery
  3-year mortality rate for cervical neuroendocrine carcinoma
Disease-free survival | Among patients with cervical neuroendocrine carcinoma, the disease-free survival within 3 years following surgery
  3-year disease-free survival for cervical neuroendocrine carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Pengming Sun, PhD, Study Chair — Fujian Maternity and Child Health Hospital, Affiliated Hospital of Fujian Medical University
Locations (9):
- China (9):
  - Fujian Maternity and Child Health Hospital, Fuzhou, Fujian
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Ningde Mindong Hospital, Ningde, Fujian
  - Putian City first Hospital, Putian, Fujian
  - The Second Affiliated Hospital of Fujian Medical University, Quanzhou, Fujian
  - Zhangzhou affiliated Hospital of Fujian Medical University, Zhangzhou, Fujian
  - Maternal and Child Health Hospital of Hubei Province, Wuhan, Hubei
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - Jiangxi maternal and Child Health Hospital, Nanchang, Jiangxi